CLINICAL TRIAL: NCT03353636
Title: A Randomized, Double-blind, Placebo-controlled, Crossover Trial to Compare the Bioavailability of Magnesium From Magnesium Carbonate Powder With Three Marketed Magnesium Supplements
Brief Title: Bioavailability of Magnesium Supplements
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Natural Calm Canada (Industry)
Collaborators: Nutrasource Pharmaceutical and Nutraceutical Services, Inc. (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: TOPN-1501
Record Dates: First submitted 2017-11-21; First posted 2017-11-27 (Actual); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Healthy; Magnesium Deficiency
MeSH Terms: conditions — Magnesium Deficiency | interventions — Magnesium

STUDY DESIGN:
Intervention Model Description: Five period crossover study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Natural Calm Magnesium (Experimental): 150mg elemental magnesium in a single oral dose
  Interventions: Dietary Supplement: Magnesium
- Magnesium Bis-glycinate (Active Comparator): 150mg elemental magnesium in a single oral dose
  Interventions: Dietary Supplement: Magnesium
- MAGSmart (Active Comparator): 150mg elemental magnesium in a single oral dose
  Interventions: Dietary Supplement: Magnesium
- Magnesium citrate (Active Comparator): 150mg elemental magnesium in a single oral dose
  Interventions: Dietary Supplement: Magnesium
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Magnesium — 150mg elemental magnesium
  Arms: MAGSmart; Magnesium Bis-glycinate; Magnesium citrate; Natural Calm Magnesium
Dietary Supplement: Placebo — Rice flour
  Arms: Placebo

SUMMARY:
The primary objective of this clinical trial is to demonstrate the superiority of Natural Calm magnesium powder with respect to absorption when compared to three marketed forms of magnesium (two magnesium bisglycinate powders and magnesium citrate capsules). The primary endpoints were serum magnesium AUC (0-8h) and urine magnesium AUC (0-8h) after a single dose of 150 mg elemental magnesium.

ELIGIBILITY:
Inclusion Criteria:

* Female 35-65 years of age
* Post-menopausal (greater than 1 year since last menses)
* Healthy as determined by blood chemistry, hematology, urinalysis and past medical history
* BMI 18-27.5 kg/m2
* Normal blood magnesium between 0.65 and 1.05mmol/L
* Normal urinary creatinine clearance 1.18 - 2.18mL/s
* Non-smoker or ex-smoker for greater than 6 months
* Agrees to maintain current dietary and physical activity habits for the duration of the study period except as instructed during run-in periods and on test days
* Willing and able to provide voluntary, written, informed consent

Exclusion Criteria:

* Woman who is peri-menopausal, premenopausal, pregnant, breastfeeding, or planning to become pregnant during the course of the trial
* Significant cardiac history defined as a history of myocardial infarction (MI); coronary angioplasty or bypass graft(s); valvular disease or repair; unstable angina pectoris; trans ischemic attack (TIA); cerebrovascular accidents (CVA); congestive heart failure; or coronary artery disease (CAD)
* Uncontrolled hypertension defined as untreated systolic blood pressure > 160 mmHg and/or diastolic blood pressure > 100 mmHg
* Uncontrolled diabetes defined as fasting blood glucose > 7 mmol/L
* Treated or untreated thyroid disorders
* History of renal and/or liver disease
* History of clinically significant gastrointestinal pathology (e.g. chronic diarrhea, inflammatory bowel disease) unresolved gastrointestinal symptoms (e. g. diarrhea, vomiting) or other diseases known to interfere with absorption, distribution, metabolism or excretion of the IP or comparators
* History of (in previous 5 years), or currently being treated for cancer (excluding basal cell skin carcinoma)
* Unstable psychiatric disorder
* Acute illness, as judged by the Investigator, within 2 weeks of the first treatment period (Visit 3a)
* Immunocompromised individuals such as participants that have undergone organ transplantation or participants diagnosed with human immunodeficiency virus (HIV)
* History of hemoglobinopathies such as sickle cell anemia or thalassemia, sideroblastic anemia
* Significant abnormal liver function as defined as AST and/or ALT > 2x the upper limit of normal (ULN), and/or bilirubin > 2 x the ULN
* Serum creatinine > 95 umol/L
* Anemia of any etiology defined as hemoglobin < 110 g/L for females
* Use of anticoagulants, statins, or any other medication for the treatment of hypercholesterolemia and/or hypertension
* Use of prescribed medication or over the counter supplements for weight loss
* Use of acute medication, including antacids, within 72 hours of study supplement dose
* Use of over the counter or prescription products containing magnesium and/or calcium (e.g. multivitamins, calcium carbonate, etc.) within 2 weeks of screening (Visit 1a)
* Use of medications known to interact or interfere with magnesium absorption (See section 3.8.2)
* Use of nicotine-containing products in any form (eg, chewing tobacco, gum, patch) within 30 days of the first test period (Visit 3a)
* Use of caffeine supplements
* Consumption of more than 50g of chocolate per day
* Excessive consumption of caffeinated beverages (e.g. >2 cups of any combination of tea, coffee, energy drinks, caffeinated soda, etc. per day) or participants who experience caffeine withdrawal headaches
* Allergy or sensitivity to study supplement ingredients
* Food allergies or sensitivities to any of the foods outlined in Appendix 2.
* Vegan or vegetarian
* Recent change in weight (up or down more than 10 % of usual body weight, within the past year)
* Participants who work, evening or night shifts
* Donation or loss of whole blood prior to the administration of the study product as follows: 50-300 mL of whole blood within 30 days, 301-500 mL of whole blood within 45 days or more than 500 mL within 56 days prior to the administration of the IP or comparators
* Presence or history (past 6 months) of alcohol or drug abuse; alcohol use of >2 standard alcoholic drinks per day
* Participant is unwilling or unable to abide by the requirements of the protocol
* Any condition that would interfere with the participant's ability to comply with study instructions, might confound the interpretation of the study, or put the participant at risk
* Participant has taken an investigational medicine or has participated in a research study within 30 days prior to the run-in period (Visit 2a)

Ages: 35 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-06-27 (Actual); Primary Completion 2017-02-03 (Actual); Study Completion 2017-02-06 (Actual)

PRIMARY OUTCOMES:
Serum Magnesium AUC | 0-8 hours
  serum magnesium area under the concentration time curve
Urinary Magnesium AUC | 0-12 hours
  urine magnesium area under the concentration time curve

SECONDARY OUTCOMES:
Serum Magnesium AUC | 0-12 hours
  serum magnesium area under the concentration time curve
Urine Magnesium AUC | 0-12 hours
  urine magnesium area under the concentration time curve
Urine Magnesium AUC | 0-24 hours
  urine magnesium area under the concentration time curve
Serum Magnesium Cmax | 12 hours
  serum magnesium maximum concentration
Serum Magnesium Tmax | 12 hours
  serum magnesium time of maximum concentration
Urine Magnesium Cmax | 24 hours
  urine magnesium maximum concentration
Urine Magnesium Tmax | 24 hours
  urine magnesium time of maximum concentration
Total urine magnesium | 24 hours
  total amount of magnesium collected in urine over 24h bioavailability period

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Bier, MD, Principal Investigator — Nutrasource Pharmaceutical and Nutraceutical Services, Inc.
Locations (1):
- Nutrasource, Guelph, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No